CLINICAL TRIAL: NCT05497011
Title: A Randomized Controlled Study to Evaluate the Safety and Efficacy of Pressure-controlled Intermittent Coronary Sinus Occlusion (PiCSO) in Anterior STEMI Patients With TIMI 0-2 at Presentation.
Brief Title: A Study to Evaluate the Safety and Efficacy of PiCSO in Anterior STEMI Patients
Acronym: PiCSO-AMI-II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of financing
Sponsor: Miracor Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIR-CIP 0003
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Anterior Wall Myocardial Infarction
Keywords: PiCSO; PiCSO Impulse System
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Anterior Wall Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, controlled, parallel-groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control (No Intervention): This is the actual control group receiving conventional therapy, ie. percutaneous coronary intervention.
- PiCSO (Experimental): This arm will be treated with Pressure controlled intermittent Coronary Sinus Occlusion (PiCSO) in addition to conventional therapy (percutaneous coronary intervention).
  Interventions: Device: PiCSO Impulse System

INTERVENTIONS:
Device: PiCSO Impulse System — After blood flow restoration, the subjects meeting all eligibility criteria will be enrolled into the study and randomized either to PiCSO Group or Control Group. If the subject is randomized to PiCSO Group, the coronary sinus (CS) will be cannulated through the femoral vein and the PiCSO Impulse Catheter will be placed in the CS. Once PiCSO Impulse Catheter is placed into CS, PiCSO treatment is started followed by stenting. The physician shall target a PiCSO treatment of 45 minutes whereas the treatment should be continued during and post stent insertion. At the end of the PiCSO treatment, the PiCSO Impulse Console is stopped and the PiCSO Impulse Catheter is removed.
  Arms: PiCSO

SUMMARY:
The objective of this study is to assess the safety and efficacy of Pressure-controlled intermittent Coronary Sinus Occlusion (PiCSO) as adjunct to percutaneous coronary intervention (PCI) compared to PCI in the setting of acute anterior ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
This is a multicenter, randomized (2 PiCSO :1 Control), controlled, pivotal study to evaluate safety and feasibility of Pressure-controlled intermittent Coronary Sinus Occlusion (PiCSO) therapy in patients with acute anterior ST-segment elevation myocardial infarction (STEMI), presenting with thrombolysis in myocardial infarction (TIMI) 0, 1, or 2 and symptom duration ≤ 12 hours treated adjunct to PCI compared to standard PCI. Patients with an ST-segment elevated anterior infarct eligible for PCI will be invited to participate in the PiCSO-AMI-II anterior STEMI study. After consent as per approved ethics committee requirements, baseline assessments will be performed. PCI of the culprit vessel should be performed per standard practices. After TIMI flow restoration, the subjects meeting all eligibility criteria will be enrolled into the study and randomized either to PiCSO Group or Control Group. If the subject is randomized to PiCSO Group, the coronary sinus (CS) will be cannulated through the femoral vein and the PiCSO Impulse Catheter will be placed in the CS. In the event the PiCSO Impulse Catheter cannot be placed in the CS within 30 minutes, the physician should proceed with the regular PCI and the PiCSO treatment will be considered a failure. Once PiCSO Impulse Catheter is placed into CS, PiCSO treatment is started followed by stenting. The physician shall target a PiCSO treatment of 45 minutes whereas the treatment should be continued during and post stent insertion. At the end of the PiCSO treatment, the PiCSO Impulse Console is stopped and the PiCSO Impulse Catheter is removed. The patient is seen at 5 days and 6 months for cardiovascular magnetic resonance imaging (CMR). Follow-up visits will take place at day 5, day 30, 6 months, 1 year, 2 years and 3 years. At every follow-up visit safety data and health status will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Culprit lesion in proximal or mid left anterior descending artery (LAD)
3. Pre-PCI TIMI flow 0, 1 or 2
4. Symptoms onset time consistent with myocardial ischemia (e.g. persistent chest pain, shortness of breath, nausea/vomiting, fatigue, palpitations or syncope) ≤ 12 h
5. Electrocardiogram (ECG) evidence of acute anterior myocardial infarction with ST-elevation ≥ 2 mm (0.2 mV) in 2 or more contiguous anterior precordial ECG leads (one of which should be V2, V3, or V4) in men or ≥ 1.5 mm (0.15 mV) in women
6. Emergent PCI will be performed according to national and local hospital guidelines
7. Consent per approved national IRB/EC specific requirements prior to the procedure.

Exclusion Criteria:

1. Patient transferred from an outside hospital where invasive coronary procedure was attempted (including diagnostic catheterization)
2. Implants or foreign bodies in the coronary sinus
3. Left main disease >= 50%
4. Need for treatment of any vessel other than the LAD (or its branches) during the index procedure or before the 5 ± 2 days study CMR.
5. Known allergy to polyurethanes, polyethylene terephthalate (PET) or stainless steel, both heparin and bivalirudin, or all of clopidogrel, ticagrelor or prasugrel that cannot be adequately pre-medicated
6. Known pregnancy or breastfeeding
7. Known large pericardial effusion or cardiac tamponade
8. Known hemodynamically relevant left to right and right to left shunt
9. Known previous myocardial infraction (MI)
10. Previous coronary artery bypass graft (CABG)
11. Known neurologic abnormality such as tumor or arteriovenous (AV) malformation, history of stroke within 6 months, any prior intracranial bleed or any permanent neurologic defect
12. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), any recent genitourinary (GU) or gastrointestinal (GI) bleed (within 3 months)
13. Administration of fibrinolytic therapy within 24 hours prior to enrollment
14. Cardiogenic shock (systolic blood pressure (SBP) < 90 mmHg), need for mechanical circulatory support, intravenous pressor or pre-randomization intubation
15. Patients with cardio-pulmonary resuscitated (CPR) cardiac arrest for more than 5 min or whom baseline neurologic status is not present
16. Patient not suitable for femoral vein access
17. Contraindication to cardiac magnetic resonance imaging CMR (e.g. claustrophobia, foreign body implants incompatible with CMR, gadolinium intolerance)
18. Active participation in another drug or device investigational study that has not reached its primary endpoint
19. Known severe kidney disease (eGFR <=30 mL/min/1.73 m2 by MDRD formula) or on hemodialysis
20. Chronic obstructive pulmonary disease (COPD) with home oxygen therapy or on chronic steroid therapy
21. Unconscious on presentation
22. Patients under judicial protection, legal guardianship or curatorship
23. Subject has other medical illness (e.g., cancer, dementia) or known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause non-compliance with the protocol, confound the data interpretation, or is associated with limited life expectancy of less than 1 year
24. Patients with definite or probable COVID-19 diagnosis > 4 weeks prior to the current MI unless they had returned to their baseline state of health after recovery from the COVID-19 illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
12% performance goal rate of PiCSO device or PiCSO procedure related adverse events reported through 30 days | 30 days post index PCI
  Primary safety endpoint is based on a 12% performance goal rate of PiCSO device or PiCSO procedure related adverse events reported through 30 days post treatment in patients randomized to PiCSO Group in which the PiCSO treatment was delivered or attempted to be delivered. These events will consist of the composite of:
  * Femoral venous access site complications:
    * Major bleed (BARC 3-5)
    * Infections requiring systemic (oral or intravenous) antibiotic treatment
    * Any femoral access site-related events requiring surgery
  * Coronary sinus dissection requiring percutaneous intervention or surgery
  * Pericardial effusion or tamponade requiring percutaneous intervention or surgery
  * Embolization or Thrombosis
  * Stroke
Difference in myocardial infarct size | 5 days post index PCI
  Difference in myocardial infarct size (extent of myocardial necrosis quantified by delayed gadolinium enhancement presented as a percentage of left ventricular (LV) mass) between the PiCSO Group and the Control Group, assessed by CMR at 5±2 days post index PCI.

SECONDARY OUTCOMES:
Major Adverse Cardiac Event (MACE) at 30 days as well as 1, 2 and 3 years post index PCI | 30 days, 1, 2 and 3 years post index PCI
  MACE at 30 days as well as 1, 2 and 3 years post index PCI
  * Cardiovascular death
  * Cardiovascular hospitalization
  * Heart failure (HF) hospitalization
  * New onset or worsening HF
Individual components of the MACE | 30 days, 1, 2 and 3 years post index PCI
  Individual components of the MACE to be evaluated at 30 days as well as 6 months and 1, 2 and 3 years post index PCI
Classification of all-cause death | 30 days, 6 months, 1, 2 and 3 years post index PCI
  Classification of all-cause death at 30 days as well as 6 months and 1, 2 and 3 years post index PCI into the following categories:
  * Cardiac cause of death
  * Non-cardiac cause of death
  * Death of Undetermined Cause
Time to death and heart failure hospitalization | 1 year post index PCI
  The hierarchical composite of time to death within 1 year, time to heart failure hospitalization within one 1-year and infarct size at assessed by CMR at 5±2 days post index PCI.
Myocardial infarct size (% of LV mass) assessed by CMR at 6 months post index PCI | 6 months post index PCI
  Myocardial infarct size (% of LV mass) assessed by CMR at 6 months post index PCI
Occurrence and extent of microvascular obstruction and hemorrhage | 5 days post index PCI
  Occurrence and extent of microvascular obstruction (MVO, % of LV mass) and hemorrhage assessed by CMR at 5 days post index PCI
Myocardial function (LVEF, LVESV, LVEDV) | 5 days and 6 months post index PCI
  Myocardial function (Left ventricular ejection fraction (LVEF), Left ventricular end-diastolic volume (LVEDV) and Left ventricular end-systolic volume (LVESV)) assessed by CMR at 5 days and 6 months post index PCI
Myocardial Salvage Index and myocardial infarct size | 5 days and 6 months post index PCI
  Myocardial Salvage Index at 5 days and 6 months post index PCI (derived from Area at Risk (AAR) assessed by CMR at 5 days and myocardial infarct size (% of LV mass) assessed by CMR at 5 days or 6 months, respectively)
ST-segment resolution | 60-90 minutes post flow restoration
  ST-segment resolution at 60-90 minutes post flow restoration
Device success and procedural success rate | Baseline (treatment day)
  Device success and procedural success rate presented as % of subjects
Changes in quality of life | 30 days, 6 months and 1, 2, 3 years post index PCI
  Changes in quality of life measured by EQ-5D at 5 days, 6 months and 1, 2, 3 years post index PCI
Utilization of health resources | 30 days, 6 months and 1, 2, 3 years post index PCI
  Assess health economics by collecting the utilization of health resources throughout the study duration

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W. Stone, Prof., Principal Investigator — Mount Sinai, New York, US